CLINICAL TRIAL: NCT01737970
Title: A Study to Correlate Ultrasound Elastography With Histopathology to Monitor the Response of Locally Advanced Breast Cancer to Neoadjuvant Chemotherapy.
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 12/SC/0170
Record Dates: First submitted 2012-11-20; First posted 2012-11-30 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
This research proposal concerns a study to monitor the effects of chemotherapy on breast cancer tumour and peritumour stromal cells using ultrasound (US) elastography (also known as strain imaging).

Many cancer treatments currently being developed are targeted; that is they exploit particular biological processes in specific cancer cell types to disrupt tumour growth. Being able to monitor the efficacy of these typically high-cost drug therapies is essential both for the best patient outcome as well as offering economical benefits to the health care system and much needed insight into future drug development.

Ultrasound provides a relatively inexpensive, non-invasive means for imaging cancers, and has been used widely in breast cancer diagnosis for many years. Its role in therapy monitoring has been suggested but has not been well explored. The purpose of this proposal is to explore this potential in more depth.

It has been identified that significant interaction takes place between tumour and stroma through all stages of tumour growth; this complex relationship is an ongoing topic of research. Fibrotic changes occur during tumour growth and are also a quintessential process of healing. Indeed, fibrosis is a common after effect to chemotherapy in many forms of cancer. Elastography is an established imaging technique (based on ultrasound or MRI) which can estimate the relative stiffness of tissues in vivo and is thus well-suited to monitor these particular biological processes.

This elucidates the main hypothesis of this project: fibrosis, cancer cell necrosis and inflammation may all contribute to a measurable response in elastography. These changes to the tissue composition can be imaged over a course of a patient's treatment to assess the response to chemo/hormonal therapy.

The ultimate project goals are to develop a clinical tool (based on ultrasound elastography) to improve treatment management in addition to offering a better biological understanding of tumour/stroma behaviour.

DETAILED DESCRIPTION:
This research proposal concerns a study to monitor the effects of chemotherapy on breast cancer tumour and peritumour stromal cells using ultrasound (US) elastography (also known as strain imaging).

Many cancer treatments currently being developed are targeted; that is they exploit particular biological processes in specific cancer cell types to disrupt tumour growth. Being able to monitor the efficacy of these typically high-cost drug therapies is essential both for the best patient outcome as well as offering economical benefits to the health care system and much needed insight into future drug development.

Ultrasound provides a relatively inexpensive, non-invasive means for imaging cancers, and has been used widely in breast cancer diagnosis for many years. Its role in therapy monitoring has been suggested but has not been well explored. The purpose of this proposal is to explore this potential in more depth.

It has been identified that significant interaction takes place between tumour and stroma through all stages of tumour growth; this complex relationship is an ongoing topic of research. Fibrotic changes occur during tumour growth and are also a quintessential process of healing. Indeed, fibrosis is a common after effect to chemotherapy in many forms of cancer. Elastography is an established imaging technique (based on ultrasound or MRI) which can estimate the relative stiffness of tissues in vivo and is thus well-suited to monitor these particular biological processes.

This elucidates the main hypothesis of this project: fibrosis, cancer cell necrosis and inflammation may all contribute to a measurable response in elastography. These changes to the tissue composition can be imaged over a course of a patient's treatment to assess the response to chemo/hormonal therapy.

The ultimate project goals are to develop a clinical tool (based on ultrasound elastography) to improve treatment management in addition to offering a better biological understanding of tumour/stroma behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Has an established diagnosis of locally advanced breast cancer.
* Aged 18 years or above.
* History of previous breast cancer does not exclude from study.
* Having neoadjuvant chemotherapy delivered in Oxford Cancer Centre.
* Good general health
* Blood tests to check suitability for the diagnostic core biopsy
* Having a localisation coil as part of routine medical care.
* Patients who are recruited into other studies can be included if there is no conflict of interest and the patient is in agreement.

Exclusion Criteria:

* Any co-morbidity that is likely to prevent regular attendance.
* Is <18 years of age or over 70 years.
* Has a movement disorder as the patient is required to lie very still for a few minutes during the scan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient will be selected from clinically diagnosed patients with breast cancer undergoing neoadjuvant chemotherapy. These women will be recruited through the Oxford University NHS Trust cancer centre and will consist primarily of women living within Oxfordshire.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The ratio of average stiffness measured within the tumour over average stiffness measured in the stroma | Patients will be followed over the course of chemotherapy treatment, an expected average of 18 weeks
  Tissue stiffness will be used to assess a patients response to chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ruth English, M.D., Principal Investigator — Oxford University NHS Trust